CLINICAL TRIAL: NCT06780436
Title: 3D Transcranial Ultrasound Brain Imaging (3D-TRUBI) Instrument for Point-of-Care Diagnosis of Intracranial Hemorrhages Caused by Traumatic Brain Injuries
Brief Title: 3D Transcranial Ultrasound Brain Imaging (3D-TRUBI) Instrument for Point-of-Care Diagnosis of Intracranial Hemorrhages
Acronym: 3D-TRUBI
Status: Active, not recruiting | Type: Observational
Sponsor: The Geneva Foundation (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C.2025.005
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Hemorrhage; Traumatic Brain Injury; Intracranial Hemorrhages; Ultrasound Exams; 3D SONOGRAPHY
Keywords: transcranial ultrasound; traumatic brain injury; intracranial hemorrhage; ultrasound
MeSH Terms: conditions — Brain Hemorrhage, Traumatic; Brain Injuries, Traumatic; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Intracranial Hemorrhage: Intracranial hemorrhage categories may include subdural hematomas, subarachnoid hemorrhages, or intraparenchymal hemorrhages.
  Interventions: Device: 3D Transcranial Ultrasound Brain Imaging
- Epidural Hematoma: Epidural hematoma group will be additionally tested to explore feasibility of scanning to this higher-acuity injury type
  Interventions: Device: 3D Transcranial Ultrasound Brain Imaging

INTERVENTIONS:
Device: 3D Transcranial Ultrasound Brain Imaging — The system implements a proprietary transcranial imaging methodology, which measures the profile of the skull bone and the speed of sound in it to accurately focus the ultrasound energy from a phased array probe through the bone in order to detect hematoma boundaries with resolution normally obtainable only through the open skull.

SUMMARY:
The primary objective of this study is to assess the safety of the 3D Transcranial Ultrasound Brain Imaging (3D TRUBI) device in Traumatic Brain Injury (TBI) patients with intracranial hemorrhage (ICH). The secondary objective is to assess the diagnostic potential of 3D TRUBI. The latter will be achieved by comparison of 3D TRUBI scans with admission head computed tomography (CT), the standard of care diagnostic modality. Demonstrating the feasibility and safety of the 3D TRUBI system is the first step toward expanding access of an alternative to CT for diagnostic imaging and triage of mass casualties of war or natural disasters in the field and in rapidly deployed medical centers or other austere environments.

DETAILED DESCRIPTION:
Eligible participants positive for intracranial hemorrhage (ICH) due to traumatic brain injury (TBI) will undergo a full scanning procedure by trained investigators. Examination with the 3D TRUBI system will involve acquisition of 16 pre-defined bilateral head points. The total time to complete the procedure is approximately 20 minutes. During the examination, feasibility and safety metrics will be collected. Additional injury data will be reviewed from participants' electronic medical record. The goal of the study is 1) to evaluate the safety of the 3D TRUBI device in the target population and 2) do demonstrate the feasibility of the device to detect ICH compared to standard medical imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Acute head injury with CT-confirmed intracranial hemorrhage
* Able to obtain written, informed consent from participant or legally authorized representative
* Able to receive intervention within 4 hours of admission head CT
* Able to feasibly receive intervention prior to neurosurgical indication

Exclusion Criteria:

* Did not receive routine head CT
* Prisoner or Wards of State
* Large or open skull wounds prohibiting ultrasound acquisition
* Received large volume fluid resuscitation (e.g. >3 units of blood product) within 2 hours of intervention
* Any prohibiting condition or contraindication for ultrasound image acquisition

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from qualifying Traumatic Brain Injuries accepted for care at Brooke Army Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intracranial Hemorrhage Detection | From enrollment to the end of data analysis (18 months)
  The primary outcome is the assessment of the feasibility of 3D-TRUBI for the detection of ICH and other traumatic brain lesions as compared to admission head CT. This is a binary parameter for each type of lesion per patient.
Evaluation of potential adverse effects | up to 48 hours after enrollment
  Participants will be evaluated for any potential adverse reactions to performance of the TRUBI exam during and after the research procedure. Twenty-four and 48-hour examination of the head are also planned to record potential adverse reactions.

SECONDARY OUTCOMES:
Morphometric comparison of 3D-TRUBI with Standard Radiology | From enrollment to end of data analysis (18 months)
  If the ICH lesion is detectable on CT, the conventional morphometric analysis of the lesion (maximum thickness, width, and length) and midline shift will be compared with morphometric analysis of the same lesions on 3D-TRUBI images. Measurements of ICH lesions by both modalities will be done in mm (millimeters), so there will be direct numerical comparisons of results using descriptive statistics, and other types of correlation and regression analyses.
Feasibility of 3D-TRUBI Assessment for Detection of Intracranial Hemorrhage | From enrollment to discharge of subject (7 days)
  To address feasibility of deployment of the 3D-TRUBI for ICH detection in the acute care setting, we will collect and analyze the time required to recruit, enroll, initiate, complete, and (where appropriate) repeat the assessment for ICH detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
To minimize risk of breaching confidentiality, individual data will not be shared with other researchers. Aggregate data may be shared upon reasonable request.

REFERENCES:
- [Background] E.R.Gr. Maev, K. Shapoori, E.V. Malyarenko, "An Ultrasonic Adaptive Beamforming Method and its Application for Transcranial Imaging", EP 3, 215, 868 B1, October 3, 2018
- [Background] D.R.Gr. Maev, K. Shapoori, E.V. Malyarenko, "An ultrasonic adaptive beamforming method and its application for transcranial imaging", US20160187473A1, June 25, 2019
- [Background] C.J. Sadler, R.Gr. Maev, E. Malyarenko, "A System to Obtain 3D Images of a Flowing Region Beneath an object using Speckle Reflections", US 9, 842, 384, December 12, 2017
- [Background] B.J. Sadler, R.Gr. Maev, E. Malyarenko, "A Method to Obtain 3D Images of a Flowing Region Beneath an object using Speckle Reflections", US 9, 613, 401, April 4, 2017
- [Background] Wydra A, Malyarenko E, Shapoori K, Maev RG. Development of a practical ultrasonic approach for simultaneous measurement of the thickness and the sound speed in human skull bones: a laboratory phantom study. Phys Med Biol. 2013 Feb 21;58(4):1083-102. doi: 10.1088/0031-9155/58/4/1083. Epub 2013 Jan 31. PMID 23363729